CLINICAL TRIAL: NCT01576016
Title: Accent Magnetic Resonance Imaging Pacemaker and Tendril Magnetic Resonance Imaging™ Lead Investigational Device Exemption Study
Brief Title: Safety and Efficacy of the Accent Magnetic Resonance Imaging™ (MRI) Pacemaker and Tendril MRI™ Lead
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 60028820
Record Dates: First submitted 2012-04-04; First posted 2012-04-12 (Estimated); Results first posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Adverse Effect of MRI on an Implanted Pacemaker Lead; Adverse Effect of MRI on an Implanted Pacemaker
Keywords: bradycardia; MRI scans
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lead Safety (Experimental): Patient implanted with an Accent MRI system to evaluate safety of the Tendril MRI lead
  Interventions: Device: Accent MRI system (lead safety)
- Accent MRI system MRI Scan Group (Experimental): Patient implanted with an Accent MRI system will receive an MRI scan to evaluate safety and efficacy of the Accent MRI system in an MRI environment
  Interventions: Device: Accent MRI system (with MRI scan)

INTERVENTIONS:
Device: Accent MRI system (lead safety) — Patients implanted with an Accent MRI system
  Other Names: Accent MRI pacemaker; Tendril MRI lead
  Arms: Lead Safety
Device: Accent MRI system (with MRI scan) — Patients implanted with an Accent MRI system will receive an MRI scan
  Other Names: Accent MRI pacemaker; Tendril MRI lead
  Arms: Accent MRI system MRI Scan Group

SUMMARY:
The MRI Study is a prospective, multi-center, clinical study designed to evaluate the safety and efficacy of the Accent MRI™ System in a patient population indicated for implant of a pacemaker within and outside of the MRI environment.

DETAILED DESCRIPTION:
The MRI Study is a prospective, multi-center, clinical study designed to evaluate the safety and efficacy of the Accent MRI System in a patient population indicated for implant of a pacemaker within and outside of the MRI environment. The study consisted of two phases, a Lead Safety Phase which evaluated the safety of the Tendril MRI lead, and an MRI Phase which evaluated the safety and efficacy of the Accent MRI pacemaker system in an MRI environment.

The safety and efficacy of the Accent MRI pacemaker and Tendril MRI lead will be evaluated as described below:

Lead Safety Safety of the Tendril MRI™ lead will be evaluated in terms of freedom from right atrial (RA) and right ventricle (RV) lead-related complications at implant to 2 months (acute timeframe), and at the 2 through the 12 month visit (chronic timeframe).

MRI Safety The safety of the Accent MRI™ system will be evaluated in terms of freedom from MRI scan related complications in the month following the MRI scan.

Lead Efficacy Efficacy of the Tendril MRI™ lead will be evaluated in terms of the change in atrial and ventricular capture and sensing thresholds before and after the MRI scan.

MRI Efficacy Efficacy of the Tendril MR lead will be evaluated in terms of the change in bipolar atrial and ventricular capture and sensing thresholds before and after the MRI scan.

Secondary Endpoints Safety Safety of the Accent MRI™ system will be evaluated in terms of freedom from system-related complications through the 12 month visit.

Efficacy Efficacy of the Tendril MRI™ lead will be evaluated in terms of the atrial and ventricular capture thresholds at the MRI Visit.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients will meet all of the following:

1. Have an approved indication per American College of Cardiology (ACC)/American Heart Association (AHA)/Heart Rhythm Society (HRS) guidelines for implantation of a pacemaker
2. Will receive a new pacemaker and lead
3. Be willing to undergo an elective MRI scan without sedation
4. Be able to provide informed consent for study participation (legal guardian is NOT acceptable)
5. Be willing and able to comply with the prescribed follow-up tests and schedule of evaluations
6. Is not contraindicated for an MRI scan (per the pre-MRI safety screening form)

Exclusion Criteria:

Patients will be excluded if they meet any of the following:

1. Are medically indicated for an MRI scan at the time of enrollment
2. Have an existing pacemaker or implantable cardioverter defibrillator (ICD). A new pacemaker and lead is required for enrollment
3. Have an existing active/inactive implanted medical device, e.g., neurostimulator, infusion pump, etc.
4. Have a non-MRI compatible device or material implanted (e.g., intracranial aneurysm clip, non-MRI compatible devices or material, metals or alloys, etc.)
5. Have a lead extender or adaptor
6. Be unable to fit in MRI bore; will come into contact with the magnet façade inside the MRI bore.
7. Have a prosthetic tricuspid heart valve
8. Are currently participating in a clinical investigation that includes an active treatment arm
9. Are allergic to dexamethasone sodium phosphate (DSP)
10. Are pregnant or planning to become pregnant during the duration of the study
11. Have a life expectancy of less than 12 months due to any condition
12. Patients with exclusion criteria required by local law (e.g., age)
13. Are unable to comply with the follow up schedule

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 950 (Actual)
Dates: Start 2012-03-30 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2018-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant Kim, Study Director — Abbott Medical Devices
Locations (70):
- United States (66):
  - University Hospital of Alabama at Birmingham, Birmingham, Alabama
  - Heart Center Research, Huntsville, Alabama
  - Arizona Arrhythmia Research Center, Phoenix, Arizona
  - Baptist Health Medical Center, Little Rock, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Mercy Hospital Northwest Arkansas, Rogers, Arkansas
  - Central Cardiology, Bakersfield, California
  - Raymond Schaerf, MD, Burbank, California
  - John Muir Medical Center, Concord, California
  - St. Jude Hospital, Fullerton, California
  - Glendale Adventist Medical Center, Glendale, California
  - Scripps Green Hospital, La Jolla, California
  - Memorial Medical Center, Modesto, California
  - Premier Cardiology, Inc / Hoag Hospital, Newport Beach, California
  - Desert Cardiology Consultants, Rancho Mirage, California
  - Mercy General Hospital, Sacramento, California
  - Sutter Memorial Hospital, Sacramento, California
  - Aurora Denver Cardiology Associates, Denver, Colorado
  - South Denver Cardiology Associates PC, Littleton, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Medical Specialists of the Palm Beaches, Atlantis, Florida
  - Watson Clinic Center, Lakeland, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Orlando Health, Orlando, Florida
  - Brevard Cardiovascular Research Associates, Rockledge, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - University of South Florida, Cardiovascular Services, Tampa, Florida
  - Athens Cardiology Group, PC, Athens, Georgia
  - Atlanta Heart Specialist, Atlanta, Georgia
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - Central Baptist Hospital, Lexington, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Spectrum Health, Grand Rapids, Michigan
  - Thoracic Cardio Healthcare Foundation, Lansing, Michigan
  - Providence Hospital, Southfield, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - St. Luke's Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Alegent Creighton Health, Omaha, Nebraska
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Mid Carolina Cardiology, Charlotte, North Carolina
  - Wake Forest University Medical Center Clinical Sciences, Winston-Salem, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Columbus Cardiovascular Associates, Columbus, Ohio
  - EMH Regional Medical Center, Elyria, Ohio
  - St. Elizabeth Health Center, Youngstown, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Oklahoma Heart Institute at Utica, Tulsa, Oklahoma
  - Abington Medical Specialists, Abington, Pennsylvania
  - Allegheny Singer Research Institute, Pittsburgh, Pennsylvania
  - Donald Guthrie Foundation for Education and Research, Sayre, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - PMG Research of Charleston, LLC, Charleston, South Carolina
  - Austin Heart, Austin, Texas
  - South Texas Cardiovascular Consultants, San Antonio, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Cardiovascular Associates, PC, Manassas, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Kitsap Cardiology Consultants, Bremerton, Washington
  - The Heart Institute at Virginia Mason, Seattle, Washington
  - Aurora Medical Group, Milwaukee, Wisconsin
- St. Andrews Hospital, Adelaide, South Australia, Australia
- Cliniques Universitaires Saint Luc, Brussels, B CAP R, Belgium
- Kuopio University Hospital, Kuopio, East Finland, Finland
- Diakonessenhuis Utrecht, Utrecht, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Lead safety phase: enrollment began on 03-30-2012 and ended on 06-18-2013; enrollment occured at 68 sites and 920 patients were enrolled.
  MRI Phase: study was approved by FDA on 03-26-2014. 255 patients were enrolled into the MRI Phase. 181 scans were completed by the 10-30-2014 cut-off date: 151 in the US, and 30 supplemental scans in Australia. The patients enrolled in the US came from the lead safety phase, the supplemental scans in Australia did not participate in lead safety phase.
Pre-assignment Details: The MRI phase was originally designed as a randomized study, with MRI and control groups, but due to challenges encountered with patient recruitment, it was later changed to a non-randomized study.
Groups:
- Lead Safety Phase: Evaluate the safety and efficacy of the St. Jude Medical Accent MRI system, which includes the Tendril MRI™ lead and Accent MRI™ pacemaker.
- MRI Safety Phase: A subset of patients enrolled in the Lead safety phase underwent an elective MRI scan to evaluate the safety and efficacy of Accent MRI system within the MRI environment.
Period: Lead Safety
Arm/Group | Lead Safety Phase | MRI Safety Phase
Started | 920 | 0
Completed | 647 | 0
Not Completed | 273 | 0
Not completed — Death | 132 | 0
Not completed — Withdrawal by Subject | 81 | 0
Not completed — System Explanted without Replacement | 24 | 0
Not completed — Physician Decision | 14 | 0
Not completed — Lost to Follow-up | 13 | 0
Not completed — Unsuccessful implant | 2 | 0
Not completed — Sponsor request | 1 | 0
Not completed — Device replaced with CRT-D | 1 | 0
Not completed — Patient on Palliative Care | 1 | 0
Not completed — Patient noncompliance | 1 | 0
Not completed — Too far from study site | 1 | 0
Not completed — System deactivated | 1 | 0
Not completed — Patient no longer followed by study PI | 1 | 0
Period: MRI Safety
Arm/Group | Lead Safety Phase | MRI Safety Phase
Started | 0 | 255 (255 enrollments includes 30 supplemental scans performed in Australia using the same scan protocol.)
Completed | 0 | 181
Not Completed | 0 | 74
Not completed — Withdrawal by Subject | 0 | 10
Not completed — Non-MRI Compatible Device or Material | 0 | 5
Not completed — Has not yet completed MRI scan | 0 | 56
Not completed — MRI scan not performed at MRI visit | 0 | 3

BASELINE CHARACTERISTICS:
Population: A subset of participants from the lead safety phase (225) were included in the "MRI Phase." 30 supplemental scans were performed in Australia for a total of 255 participants in the MRI Phase. Each Phase was analyzed separately.
Groups:
- MRI Phase: A subset of patients enrolled in the Lead safety phase (225 subjects from lead safety phase) underwent an elective MRI scan to evaluate the safety and efficacy of Accent MRI system within the MRI environment.
- Total: Total of all reporting groups
Arm/Group | Lead Safety Phase | MRI Phase | Total
Number analyzed (Participants) | 920 | 255 | 1175
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Each phase was analyzed separately.
  years
    Age - Lead Safety Phase: number analyzed (Participants) | 920 | 0 | 920
    Age - Lead Safety Phase | 73.5 (10.8) |  | 73.5 (10.8)
    Age - MRI Safety Phase: number analyzed (Participants) | 0 | 255 | 255
    Age - MRI Safety Phase |  | 70.2 (11.6) | 70.2 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Each phase was analyzed separately.
  Participants
    Sex - Lead Safety Phase: number analyzed (Participants) | 920 | 0 | 920
    Sex - Lead Safety Phase: Female | 421 |  | 421
    Sex - Lead Safety Phase: Male | 499 |  | 499
    Sex - MRI Safety Phase: number analyzed (Participants) | 0 | 255 | 255
    Sex - MRI Safety Phase: Female |  | 114 | 114
    Sex - MRI Safety Phase: Male |  | 141 | 141
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Each phase was analyzed separately Population: Analysis for lead safety and MRI safety phases was done separately.
  Participants
    Lead Safety Phase: number analyzed (Participants) | 920 | 0 | 920
    Lead Safety Phase: Hispanic or Latino | 14 | 0 | 14
    Lead Safety Phase: Not Hispanic or Latino | 904 | 0 | 904
    Lead Safety Phase: Unknown or Not Reported | 2 | 0 | 2
    MRI Safety Phase: number analyzed (Participants) | 0 | 255 | 255
    MRI Safety Phase: Hispanic or Latino | 0 | 4 | 4
    MRI Safety Phase: Not Hispanic or Latino | 0 | 251 | 251
    MRI Safety Phase: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Each phase was analyzed separately Population: Analysis for lead safety and MRI safety phases was done separately.
  Participants
    Lead Safety Phase: number analyzed (Participants) | 920 | 0 | 920
    Lead Safety Phase: American Indian or Alaska Native | 3 | 0 | 3
    Lead Safety Phase: Asian | 12 | 0 | 12
    Lead Safety Phase: Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
    Lead Safety Phase: Black or African American | 51 | 0 | 51
    Lead Safety Phase: White | 842 | 0 | 842
    Lead Safety Phase: More than one race | 0 | 0 | 0
    Lead Safety Phase: Unknown or Not Reported | 10 | 0 | 10
    MRI Safety Phase: number analyzed (Participants) | 0 | 255 | 255
    MRI Safety Phase: American Indian or Alaska Native | 0 | 1 | 1
    MRI Safety Phase: Asian | 0 | 2 | 2
    MRI Safety Phase: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    MRI Safety Phase: Black or African American | 0 | 20 | 20
    MRI Safety Phase: White | 0 | 229 | 229
    MRI Safety Phase: More than one race | 0 | 0 | 0
    MRI Safety Phase: Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants] — Region of enrollment lead safety phase. Each phase of the study was analyzed separately Population: Region of enrollment for lead safety phase only. Each phase of the study was analyzed separately
  participants
    United States: number analyzed (Participants) | 920 | 0 | 920
    United States | 920 |  | 920
Region of Enrollment [Number; unit: participants] — Region of enrollment MRI safety phase. Each phase of the study was analyzed separately Population: Region of enrollment for MRI safety phase only. Each phase of the study was analyzed separately
  participants
    United States: number analyzed (Participants) | 0 | 225 | 225
    United States |  | 225 | 225
    Australia: number analyzed (Participants) | 0 | 30 | 30
    Australia |  | 30 | 30
Primary Indication for Pacemaker Implant [Count of Participants; unit: Participants] — Population: Each phase was analyzed separately.
  Participants
    Lead Safety Phase: number analyzed (Participants) | 920 | 0 | 920
    Lead Safety Phase: AV block | 246 |  | 246
    Lead Safety Phase: Other | 19 |  | 19
    Lead Safety Phase: Pacemaker Generator Change | 2 |  | 2
    Lead Safety Phase: Prevention/Termination Of Tachyarrhythmias By Paci | 13 |  | 13
    Lead Safety Phase: Sinus Node Dysfunction | 581 |  | 581
    Lead Safety Phase: Syncope | 59 |  | 59
    MRI Safety Phase: number analyzed (Participants) | 0 | 255 | 255
    MRI Safety Phase: AV block |  | 65 | 65
    MRI Safety Phase: Other |  | 7 | 7
    MRI Safety Phase: Pacemaker Generator Change |  | 1 | 1
    MRI Safety Phase: Prevention/Termination Of Tachyarrhythmias By Paci |  | 5 | 5
    MRI Safety Phase: Sinus Node Dysfunction |  | 159 | 159
    MRI Safety Phase: Syncope |  | 18 | 18
Cardiovascular History [Count of Participants; unit: Participants] — Population: Each phase was analyzed separately
  Participants
    Lead Safety Phase: number analyzed (Participants) | 920 | 0 | 920
    Lead Safety Phase: Coronary Artery Disease | 338 |  | 338
    Lead Safety Phase: Myocardial Infarction | 119 |  | 119
    Lead Safety Phase: Unstable Angina | 73 |  | 73
    Lead Safety Phase: None | 390 |  | 390
    MRI Safety Phase: number analyzed (Participants) | 0 | 255 | 255
    MRI Safety Phase: Coronary Artery Disease |  | 35 | 35
    MRI Safety Phase: Myocardial Infarction |  | 5 | 5
    MRI Safety Phase: Unstable Angina |  | 6 | 6
    MRI Safety Phase: None |  | 209 | 209
Prior Cardiac Interventions [Count of Participants; unit: Participants] — Population: Each phase was analyzed separately
  Participants
    Lead Safety Phase: number analyzed (Participants) | 920 | 0 | 920
    Lead Safety Phase: Ablation | 100 |  | 100
    Lead Safety Phase: Coronary Artery Bypass Graft | 130 |  | 130
    Lead Safety Phase: PTCA/Stents/Atherectomy | 152 |  | 152
    Lead Safety Phase: None | 538 |  | 538
    MRI Safety Phase: number analyzed (Participants) | 0 | 255 | 255
    MRI Safety Phase: Ablation |  | 38 | 38
    MRI Safety Phase: Coronary Artery Bypass Graft |  | 2 | 2
    MRI Safety Phase: PTCA/Stents/Atherectomy |  | 8 | 8
    MRI Safety Phase: None |  | 207 | 207
Non-Ventricular Arrhythmia History [Number; unit: participants] — Each phase was analyzed separately
  participants
    Paroxysmal AF - lead safety | 316 | 0 | 316
    Paroxysmal AF - MRI safety | 0 | 79 | 79
    Permanent AF - lead safety | 63 | 0 | 63
    Permanent AF - MRI safety | 0 | 16 | 16
    Persistent AF - lead safety | 100 | 0 | 100
    Persistent AF - MRI safety | 0 | 23 | 23
    Atrial Flutter - lead safety | 123 | 0 | 123
    Atrial Flutter - MRI safety | 0 | 39 | 39
    Atrial Tachycardia - lead safety | 41 | 0 | 41
    Atrial Tachycardia - MRI safety | 0 | 16 | 16
    Supra Ventricular - lead safety | 55 | 0 | 55
    Supra Ventricular - MRI safety | 0 | 10 | 10
    None - lead safety | 370 | 0 | 370
    None - MRI safety | 0 | 111 | 111

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Right Atrial (RA) Lead-related Complications in the Acute Period
Description: Percentage of patients who do not have RA lead-related complications from implant through the 2 month study visit
Time Frame: Implant through 2 months
Population: 99 of the 920 enrolled subjects had no RA lead and hence did not contribute any data towards this endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Lead Safety Phase
Number analyzed (Participants) | 821
percentage of subjects | 97.2 [95.81 to 98.13]

2. Primary Outcome: Freedom From Right Ventricular (RV) Lead-related Complications in the Acute Time Period
Description: Percentage of patients who do not have RV lead-related complications from implant through the 2 month study visit
Time Frame: Implant through 2 months
Population: one of 920 enrolled subjects did not have an RV lead implanted.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Lead Safety Phase
Number analyzed (Participants) | 919
percentage of subjects | 98.45 [96.81 to 99.25]

3. Primary Outcome: Freedom From RA Related Complications in the Chronic Period
Description: Percentage of patients who do not have RA lead-related complications from the 2 month through the 12 month study visit
Time Frame: 2 months through 12 months
Population: Data from 114 subjects were unavailable for this endpoint analysis due to the following reasons: no RA lead: 99; death: 8; unsuccessful implant: 2; withdrawal:5.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Lead Safety Phase
Number analyzed (Participants) | 806
percentage of subjects | 98.82 [97.04 to 99.53]

4. Primary Outcome: Freedom From Right Ventricular Lead Related Complications in the Chronic Period
Description: Percentage of patients who do not have RV lead-related complications from the 2 month through the 12 month study visit
Time Frame: 2 months through 12 months
Population: Data from 18 subjects were unavailable for this endpoint analysis due to the following reasons: no RV lead: 1; death: 9; unsuccessful implant: 2; withdrawal: 6.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Lead Safety Phase
Number analyzed (Participants) | 902
percentage of subjects | 100 [100.00 to 100.00]

5. Primary Outcome: Freedom From MRI Scan-related Complications
Description: Percentage of patients who do not have MRI-related complications from the MRI scan visit to the 1 month post MRI scan visit
Time Frame: MRI Scan visit through 1 month after MRI scan visit
Population: 151 of the 255 patients enrolled received an MRI scan. An additional 30 scans were performed using an identical scan protocol implemented in this study, for a total of 181 patients who underwent an MRI scan.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- MRI Safety Phase: Evaluate the safety and efficacy of the St. Jude Medical Brady MRI system, which includes the Tendril MRI™ lead and Accent MRI™ pacemaker, within the MRI environment.
Arm/Group | MRI Safety Phase
Number analyzed (Participants) | 181
percentage of subjects | 100 [98.37 to 100.00]

6. Primary Outcome: Change in Atrial Capture Threshold From Pre to Post MRI Scan
Description: Percentage of patients with an increase in RA capture thresholds of <= 0.5 V, at a pulse width of 0.5 ms .
Time Frame: MRI Scan visit to 1 month after MRI scan visit
Population: 37 of the 181 subjects that underwent a MRI scan did not have RA capture threshold data at 1-month post scan; no RA lead: 10; RA lead off: 3; atrial fibrillation (AF/AFl) during measurement: 10; 1-month visit not completed: 14.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- MRI Efficacy Phase: Evaluate the efficacy of the St. Jude Medical Brady MRI system, which includes the Tendril MRI™ lead and Accent MRI™ pacemaker, within the MRI environment.
Arm/Group | MRI Efficacy Phase
Number analyzed (Participants) | 144
percentage of subjects | 100 [97.47 to 100.00]

7. Primary Outcome: Change in Ventricular Capture Threshold Pre to Post MRI Scan
Description: Percentage of patients with an increase in RV capture thresholds of <=0.5V, at a pulse width of 0.5 ms.
Time Frame: MRI Scan visit to 1 month after MRI scan visit
Population: 167 of the 181 subjects with an MRI scan had completed the 1-month post MRI visit. Data from 167 subjects was available for this analysis; 13 subjects had not completed 1 month follow-up, 1 subject had RV capture threshold missing or not done.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | MRI Efficacy Phase
Number analyzed (Participants) | 167
percentage of subjects | 100 [97.82 to 100.00]

8. Primary Outcome: Change in Atrial Sense Amplitude
Description: Percentage of patients with a reduction in RA sense amplitude <=50 % and sense amplitude >=1.5 mV.
Time Frame: MRI Scan visit to 1 month after MRI scan visit
Population: 60 of the 181 subjects that underwent an MRI scan did not have RA sense amplitude data: no RA lead: 10; RA lead off: 3; AF/AFl/ heart rate< 30 bpm/ no P-wave during measurement: 11; P-wave < 1.5 mV: 23; 1-month visit not yet completed: 12; AF/AFl during 1-month measurement: 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | MRI Efficacy Phase
Number analyzed (Participants) | 121
percentage of subjects | 92.56 [86.35 to 96.54]

9. Primary Outcome: Change in Ventricular Sense Amplitude
Description: Percentage of patients with an reduction in RV sense amplitude <=50% and sense amplitude >=5 mV.
Time Frame: MRI Scan visit to 1 month after the MRI Scan visit
Population: 47 of 181 subjects that underwent an MRI scan did not have RV sense amplitude: no R-wave/HR < 30 beats per minute (BPM): 18; R-wave amplitude < 5 mV: 18; one-month visit not completed: 11. 134 subjects were available for evaluation of endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | MRI Efficacy Phase
Number analyzed (Participants) | 134
percentage of subjects | 97.76 [93.6 to 99.5]

10. Secondary Outcome: Freedom From System-related Complications
Description: Percentage of patients who do not have system-related complications from implant through the 12 month study visit
Time Frame: Implant through 12 months
Population: All subjects enrolled in the lead-safety arm.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Lead Safety Phase
Number analyzed (Participants) | 920
percentage of subjects | 94.64 [92.76 to 96.05]

11. Secondary Outcome: Atrial Capture Threshold at the MRI Visit
Description: Percentage of patients with RA capture threshold ≤2.0 volts (V) at the MRI visit
Time Frame: MRI Scan visit (approx 3 months post implant)
Population: 23 of the 181 subjects that underwent an MRI scan did not have RA capture threshold for the MRI scan visit: no RA lead: 10; RA lead off: 3; AF/AFl during measurement: 10.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- MRI Efficacy Phase: Evaluate the efficacy of the St. Jude Medical Accent MRI system, which includes the Tendril MRI™ lead and Accent MRI™ pacemaker, within the MRI environment.
Arm/Group | MRI Efficacy Phase
Number analyzed (Participants) | 158
percentage of subjects | 100.00 [97.69 to 100.00]

12. Secondary Outcome: Ventricular Capture Threshold at the MRI Visit
Description: Percentage of patients with RV capture threshold ≤2.0 V at the MRI visit
Time Frame: MRI Scan visit (approx 3 months post implant)
Population: All subjects that underwent a MRI scan had ventricular capture threshold data available.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | MRI Efficacy Phase
Number analyzed (Participants) | 181
percentage of subjects | 100.00 [97.98 to 100.00]

ADVERSE EVENTS:
Time Frame: 5 years
Description: Adverse events (AEs) are classified as complications, observations, or other reported events. An independent, Clinical Events Committee, adjudicated all adverse events reported during the MRI Study.
  Complications: AEs that require invasive intervention.
  Observations: AEs that can be managed without invasive intervention.
  Other Reported Events (ORE): Any other clinical event, which is not caused/associated with the study system component(s) and/or defined as an AE.
Groups:
- MRI Phase: Evaluate the safety and efficacy of the St. Jude Medical Accent MRI system, which includes the Tendril MRI™ lead and Accent MRI™ pacemaker, within the MRI environment.
Arm/Group | Lead Safety Phase | MRI Phase
All-Cause Mortality (participants affected / at risk) | 132/920 | 0/255
Serious Adverse Events (participants affected / at risk) | 70/920 | 0/255
Other Adverse Events (participants affected / at risk) | 60/920 | 1/255
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead Safety Phase (N=920) | MRI Phase (N=255)
RA Lead Related: Lead Dislodgement or Migration (Product Issues) | 24 (26) | 0 (0)
RA Lead Related: Elevated Pacing Thresholds (Product Issues) | 2 (2) | 0 (0)
RA Lead Related: Cardiac Perforation (Product Issues) | 1 (1) | 0 (0)
RA Lead Related: Lead Fracture (Product Issues) | 1 (1) | 0 (0)
RA Lead Related: Undersensing (Product Issues) | 1 (1) | 0 (0)
RV Lead Related: Lead Dislodgement or Migration (Product Issues) | 7 (7) | 0 (0)
RV Lead Related: Elevated Pacing Thresholds (Product Issues) | 1 (1) | 0 (0)
VR Lead Related: Lead Fracture (Product Issues) | 1 (1) | 0 (0)
RV Lead Related: Loss of Capture (Product Issues) | 1 (1) | 0 (0)
RV Lead Related: Extracardiac Stimulation (Product Issues) | 1 (1) | 0 (0)
RV Lead Related: Twiddler's Syndrome (General disorders) | 1 (1) | 0 (0)
Pacemaker Related: Device Connectivity Issue (Product Issues) | 1 (1) | 0 (0)
Pacemaker Related: Early Battery Depletion (Product Issues) | 1 (1) | 0 (0)
System Related: Cardiac Tamponade (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
System Related: Decompensated HF (Cardiac disorders) | 2 (2) | 0 (0)
System Related: Infection (Infections and infestations) | 2 (2) | 0 (0)
System Related: Pacemaker Induced Cardiomyopathy (Cardiac disorders) | 2 (2) | 0 (0)
System Related: Cardiac Perforation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
System Related: Pacemaker system relocation to right side (General disorders) | 1 (1) | 0 (0)
System Related: Pericardial Effusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedure Related: Pneumothorax (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Procedure Related: Infection (Infections and infestations) | 3 (3) | 0 (0)
Procedure Related: Bleeding/Hematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedure Related: Pocket Site/Incision Pain Lasting Greater Than 72 Hours Post Implant (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedure Related: Insufficient Slack in Lead (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Procedure Related: Device Migration (Product Issues) | 1 (1) | 0 (0)
Procedure Related: Hemoptysis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedure Related: Hemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedure Related: Pericardial Effusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedure Related: Stenosis of The Left Subclavian Vein (Vascular disorders) | 1 (1) | 0 (0)
Procedure Related: Thrombo-Embolic Event (Vascular disorders) | 1 (1) | 0 (0)
Procedure Related: Wound Dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead Safety Phase (N=920) | MRI Phase (N=255)
RA Lead Related: Oversensing (Product Issues) | 7 (7) | 0 (0)
Pacemaker Related: Pacemaker Mediated Tachycardia (General disorders) | 30 (32) | 1 (1)
Procedure Related: Bleeding/Hematoma (Injury, poisoning and procedural complications) | 9 (9) | 0 (0)
Procedure Related: Pneumothorax (Injury, poisoning and procedural complications) | 7 (7) | 0 (0)
Procedure Related: Thrombo-Embolic Event (Vascular disorders) | 7 (7) | 0 (0)
ORE: Atrial Arrhythmia (Cardiac disorders) | 46 (56) | 0 (0)
ORE: Decompensated HF (Cardiac disorders) | 17 (22) | 0 (0)
ORE: Ventricular Arrhythmia (Cardiac disorders) | 14 (16) | 0 (0)
ORE: Chest Pain (Cardiac disorders) | 7 (8) | 0 (0)
ORE: Cerebrovascular Accident (Vascular disorders) | 8 (9) | 0 (0)
ORE: Angina (Cardiac disorders) | 7 (10) | 0 (0)
ORE: Syncope (Cardiac disorders) | 5 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2014-07-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT01576016/Prot_SAP_ICF_000.pdf